CLINICAL TRIAL: NCT03811795
Title: Cryoballoon vs. Rhythmia Guided Ablation for Recurrent Atrial Fibrillation Following Initial Cryoballoon Pulmonary Vein Isolation
Brief Title: Cryoballoon vs. Rhythmia Guided Ablation for Recurrent AFib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABCRYO1786
Record Dates: First submitted 2018-12-20; First posted 2019-01-22 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The study is a randomized, prospective multicenter pilot study to assess the utility and efficacy of high-density mapping with the Rhythmia mapping system to guide PV re-isolation in subjects with recurrent AF after an initial cryoballoon PVI compared to repeat cryoballoon PVI.
  After obtaining informed consent to participate in the study, subjects will undergo baseline data collection. Subjects will then be randomized to undergo repeat PVI with either cryoballoon ablation or repeat PVI with an IntellaNav Open-Irrigated or other approved ablation catheters for atrial fibrillation under guidance of the Rhythmia mapping system and IntellaMap Orion mapping catheter. The performance of repeat AF ablation, use either the cryoballoon or Rhythmia mapping system, mapping catheter, and ablation catheters are in accordance with standard clinical indications and practice, regardless of participation in the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1-Repeat Cryoballoon Ablation (Other): Subjects will be randomized to repeat cryoballoon ablation.
  Interventions: Other: ECG monitoring with a Kardia Mobile monitor
- Arm 2-Radiofrequency Ablation (Other): Participants will have radiofrequency ablation guided by high-fidelity mapping (Rhythmia) following an initial cryoballoon ablation.
  Interventions: Other: ECG monitoring with a Kardia Mobile monitor

INTERVENTIONS:
Other: ECG monitoring with a Kardia Mobile monitor — The participants in the study will undergo a total of two follow-up visits after ablation (approximately 3 and 6 months) with a 12-lead electrocardiogram at each visit. An assessment of rhythm will be performed with daily transmissions as well as subject-activated event recordings for symptoms with the Kardia Mobile smartphone based monitor. The Kardia Mobile System is an FDA-cleared, clinical grade mobile ECG monitor coupled with a smartphone app that is able to record a single-lead ECG and securely transmit the tracings to the study investigators via the Kardia Pro commercial (HIPPA compliant) remote monitoring service for clinicians.

SUMMARY:
The purpose of this research is to evaluate whether cryoballoon ablation vs. radiofrequency ablation guided by high-fidelity mapping (Rhythmia) is the best treatment strategy to perform repeat ablation for recurrent atrial fibrillation after previously having undergone cryoballoon ablation.

DETAILED DESCRIPTION:
The study is a randomized, prospective multicenter pilot study to assess the utility and efficacy of high-density mapping with the Rhythmia mapping system to guide PV re-isolation in subjects with recurrent AF after an initial cryoballoon PVI compared to repeat cryoballoon PVI.

After obtaining informed consent to participate in the study, subjects will undergo baseline data bcollection. Subjects will then be randomized to undergo repeat PVI with either cryoballoon ablation or repeat PVI with an IntellaNav Open-Irrigated or other approved ablation catheters for atrial fibrillation under guidance of the Rhythmia mapping system and IntellaMap Orion mapping catheter. The performance of repeat AF ablation, use either the cryoballoon or Rhythmia mapping system, mapping catheter, and ablation catheters are in accordance with standard clinical indications and practice, regardless of participation in the study.

The participants in the study will undergo a total of two follow-up visits after ablation (approximately 3 and 6 months) with a 12-lead electrocardiogram (ECG) at each visit. An assessment of rhythm will be performed with daily transmissions as well as subject-activated event recordings for symptoms with the Kardia Mobile (AliveCor, Mountain View, CA) smartphone based monitor. The Kardia Mobile System is an FDA-cleared, clinical grade mobile ECG monitor coupled with a smartphone app that is able to record a single-lead ECG and securely transmit the tracings to the study investigators via the Kardia Pro commercial (HIPPA compliant) remote monitoring service for clinicians. The transmissions will not be directly available to the treating electrophysiologists at each site.

At the 6 month visit, 2-weeks of continuous monitoring with a Zio XT event monitor (iRhythm, San Francisco, CA) will be performed according to standard clinical practice to evaluate for subclinical episodes of AF.

The goal of the pilot study is to enroll 50 subjects with 1:1 randomization across 3 sites in the Unites States and each subject will be followed for 6 months following ablation to evaluate for recurrence of AF. The estimated time to complete enrollment will be 3-4 months assuming enrollment of at each visit 4-5 subject per month at each site.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with paroxysmal or persistent AF undergoing repeat AF ablation as per recent HRS guidelines and standard practice;
* Individuals in whom the initial ablation approach was cryoballoon PVI at the enrolling institution more than 3 month or more prior to the anticipated repeat ablation;
* Age ≥ 18 years.

Exclusion Criteria:

* Individuals with recurrent AF who previously underwent RF-based PVI;
* Individuals with known contraindications to ablation including permanent atrial fibrillation or intolerance of anticoagulation;
* Individuals unable or not willing to complete follow-up visits and examination for the duration of the study;
* Individuals without access to smartphone or tablet compatible with the monitoring system;
* Prior valve surgery or surgical AF ablation;
* Individuals with mental or physical limitations precluding informed consent;
* Individuals currently enrolled in another investigational study or registry;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
PrimaryCryoballoon vs. Rhythmia Guided Ablation for Recurrent AFib | Six months
  The freedom from atrial fibrillation at 6 months is the primary endpoint. The presence or absence of atrial fibrillation will be assessed during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Advay Bhatt, MD, Principal Investigator — The Valley Hosptial
Locations (3):
- United States (3):
  - Iowa Heart Center, West Des Moines, Iowa
  - The Valley Hospital, Paramus, New Jersey
  - Peace Health, Springfield, Oregon